CLINICAL TRIAL: NCT06248554
Title: Adjuvant PD-1 Inhibitor for Patients With Early-stage Hepatocellular Carcinoma Following Microwave Ablation: a Prospective Cohort Study
Brief Title: Adjuvant PD-1 Inhibitor for Patients With Early-stage Hepatocellular Carcinoma Following Microwave Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Adjuvant therapy; Microwave ablation; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor adjuvant therapy group (Experimental): Received adjuvant PD-1 inhibitor 2-4 weeks after microwave surgery for a total of 9 cycles of treatment
  Interventions: Drug: PD-1 Inhibitors
- Control group (No Intervention): Receive regular monitoring and follow-up

INTERVENTIONS:
Drug: PD-1 Inhibitors — Patients in the intervention group received post-operative adjuvant PD-1 inhibitor therapy, 240 mg intravenously every three weeks for nine cycles
  Arms: PD-1 inhibitor adjuvant therapy group

SUMMARY:
For early-stage hepatocellular carcinoma, i.e. Barcelona Clinical Liver Cancer Stage 0, ablation is the standard treatment with a comparable prognosis and less risk of ablation compared with liver resection. However, ablation is demanding on the surgeon and patients often face early recurrence if ablation is not complete. Therefore, it is necessary to find reasonable adjuvant treatment to consolidate the effect of microwave therapy.

DETAILED DESCRIPTION:
For early-stage hepatocellular carcinoma, i.e. Barcelona Clinical Liver Cancer Stage 0, ablation is the standard treatment with a comparable prognosis and less risk of ablation compared with liver resection. However, ablation is demanding on the surgeon and patients often face early recurrence if ablation is not complete. Therefore, it is necessary to find reasonable adjuvant treatment to consolidate the effect of microwave therapy. There is no consensus on postoperative adjuvant therapy, especially for the management of early-stage HCC. Most scholars believe that HCC in this period does not have high-risk factors for tumor recurrence, thus neglecting the role of adjuvant therapy. Early studies have found that microwave ablation can alter the tumor microenvironment, which is conducive to the action of immune checkpoint inhibitors such as PD-1 inhibitors and even has a synergistic anti-tumor effect. We therefore designed this prospective cohort study to explore the efficacy and safety of adjuvant PD-1 inhibitors after microwave surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Pathological type is HCC, BCLC stage 0-A
* No extrahepatic HCC
* No radiographic recurrence at 2-4 weeks after ablation
* Eastern Cooperative Oncology Group (ECOG) performing status of 0-1
* Child-Pugh grade A or B and adequate hematologic and organ function

Exclusion Criteria:

* Any history of other malignant tumors or recurrent HCC
* Any preoperative treatment for HCC including local and systemic therapy
* Any acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* Any persistent serious ablation-related complications
* Esophageal and/or gastric variceal bleeding within 6 months
* Inability or refusal to comply with the treatment and monitoring
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of include in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Disease-free survival was defined as the period from inclusion in the study until tumor recurrence, death from any cause.

SECONDARY OUTCOMES:
Overall survival | From date of include in this research until the date of death from any cause, whichever came first, assessed up to 60 months
  Overall survival was defined as the period from study inclusion until death from any cause.
Adverse effects | 6 months
  Adverse reactions are defined as any reaction during treatment that is inconsistent with the purpose of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: WanGuang D Zhang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, China

IPD SHARING:
Plan to Share IPD: No